CLINICAL TRIAL: NCT02569892
Title: Non-Damaging Photothermal Therapy of Non-exudative Age Related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Bascom Palmer Eye Institute (Other)
Responsible Party: Principal Investigator, Steven R. Sanislo, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-33991
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Macular Degeneration; Retinal Drusen
MeSH Terms: conditions — Macular Degeneration; Retinal Drusen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Arm (Experimental): Participants receive treatment with sub-threshold macular laser photocoagulation
  Interventions: Device: Pascal Retinal Laser Photocoagulator
- Sham Laser Arm (Sham Comparator): Participants receive sham treatment with sub-threshold macular laser photocoagulation (with power setting at zero)
  Interventions: Device: Pascal Retinal Laser Photocoagulator

INTERVENTIONS:
Device: Pascal Retinal Laser Photocoagulator — Sub-threshold macular laser treatment with Pascal laser Endpoint Management System

SUMMARY:
This is a randomized controlled study of non-damaging photothermal macular grid laser versus sham laser therapy in patients with dry age-related macular degeneration (AMD) and large high-risk drusen. The goal of the study is to determine if this treatment will reduce macular drusen volume and also whether this might improve visual acuity or reduce the risk of conversion to advanced age-related macular degeneration defined as development of choroidal neovascularization or geographic atrophy.

ELIGIBILITY:
Inclusion Criteria

1. Older than 60 years of age.
2. Male or female patients with nonexudative AMD with a drusen volume of of at least 0.03mm3 in the central 3mm circle
3. Adequate pupil dilatation and clear media to perform colour, red-free imaging and fundus fluorescein angiography, fundus autofluorescence imaging and OCT.
4. Able to give an informed consent.

Exclusion Criteria:

1. Presence of signs of advanced AMD, such as CNV, haemorrhages or macular atrophy based on OCT and fundus autofluorescence photography (FAF).
2. Previous macular laser treatment.
3. Any previous ocular condition that may be associated with a risk of developing macular oedema.
4. Vitreomacular traction determined clinically and /or by OCT, which in the opinion of the investigator, contributes to the macular oedema (associated or causing a detachment of the fovea).
5. Presence of other macular disease such as epiretinal membrane, macular telangiectasia.
6. Important known allergies to sodium fluorescein dye used in angiography.
7. Ocular or periocular infections.
8. Planned intra-ocular surgery within one year.
9. Patient is unavailable for follow-up visits.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sanislo, MD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from January 2016 until May 2018, at which time interim analysis revealed futility.
Pre-assignment Details: 19 participants signed informed consent; 2 participants failed screening, and 17 participants started the study. Participants may have contributed one or both eyes to the study. If both eyes were enrolled the first eye would be randomly assigned to treatment or sham, and the fellow eye would be assigned to the opposite treatment arm. Participants who contributed more than one eye are counted in more than one reporting group.
Units Other Than Participants: Eyes
Groups:
- Sub-threshold Macular Laser Photocoagulation: Participants that receive treatment with sub-threshold macular laser photocoagulation
- Sham Laser: Participants that receive sham treatment with sub-threshold macular laser photocoagulation (with power setting at zero)
Period: Overall Study
Arm/Group | Sub-threshold Macular Laser Photocoagulation | Sham Laser
Started | 10; 10 Eyes | 9; 9 Eyes
Completed | 10; 10 Eyes | 8; 8 Eyes
Not Completed | 0; 0 Eyes | 1; 1 Eyes

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- All Participants: Participants receive sub-threshold macular laser photocoagulation and/or sham treatment with power setting at zero
Arm/Group | All Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Macular Drusen Volume
Description: Mean change in macular drusen volume as measured on high-resolution spectral domain ocular coherence tomography (SD-OCT)
Time Frame: baseline, 6, 12, and 24 months
Population: Participants who contributed more than one eye are counted in more than one reporting group. Data for the participant who did not complete the study are included using the Last Observation Carried Forward (LOCF) method.
Measure: Median (Inter-Quartile Range); unit: mm^3
Units Other Than Participants: Eyes
Arm/Group | Sub-threshold Macular Laser Photocoagulation | Sham Laser
Number analyzed (Participants) | 10 | 9
Number analyzed (Eyes) | 10 | 9
mm^3
  Baseline volume | 0.05 [0.05 to 0.14] | 0.11 [0.07 to 0.13]
  6 month change | 20.0 [6.04 to 33.30] | 9.0 [-55.50 to 25.00]
  12 month change | 42.2 [25.00 to 55.01] | 27.2 [-85.70 to 46.20]
  24 month change | 80.0 [34.75 to 135.00] | -4.5 [-85.70 to 81.80]

2. Secondary Outcome: Change in Visual Acuity
Description: Mean change in best-corrected visual acuity as measured using early treatment diabetic retinopathy study (ETDRS) chart - average number of letters seen on chart
Time Frame: baseline, 6, 12, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Units Other Than Participants: Eyes
Arm/Group | Sub-threshold Macular Laser Photocoagulation | Sham Laser
Number analyzed (Participants) | 10 | 9
Number analyzed (Eyes) | 10 | 9
Letters
  Baseline vision | 81.7 (8.60) | 79.4 (5.19)
  6 month change | -0.7 (4.24) | -3.4 (4.67)
  12 month change | -2.7 (324) | -0.9 (3.95)
  24 month change | -3.6 (6.10) | -6.3 (6.96)

3. Secondary Outcome: Development of Geographic Atrophy (GA) or Choroidal Neovascularization (CNV)
Description: Count of eyes that develop geographic atrophy or choroidal neovascularization by 24 months.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Sub-threshold Macular Laser Photocoagulation | Sham Laser
Number analyzed (Participants) | 10 | 9
Number analyzed (Eyes) | 10 | 9
Eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Per protocol, only adverse events related to treatment were collected. Participants who contributed more than one eye are counted in more than one reporting group.
Arm/Group | Sub-threshold Macular Laser Photocoagulation | Sham Laser
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub-threshold Macular Laser Photocoagulation (N=10) | Sham Laser (N=9)
mild supra-threshold laser burns (Eye disorders) | 1 (1) | 0 (0) — Laser burns in this study were to be sub-threshold (non-visible).

LIMITATIONS AND CAVEATS:
This study did not meet enrollment goal of 60 study eyes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02569892/Prot_SAP_000.pdf